CLINICAL TRIAL: NCT06844526
Title: Comparative Effects of Core Stability Exercises Versus Hopping Exercises on Trunk Stability and Balance Among Kabaddi Athletes
Brief Title: Comparative Effects of Core Stability Versus Hoping Exercises on Trunk Stability Among Kabaddi Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0414
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Sports Physical Therapy
Keywords: core stability exercises; hoping exercises; trunk stability and balance; kabaddi athlets

STUDY DESIGN:
Intervention Model Description: Randomized control design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hoping Exercise (Experimental)
  Interventions: Other: Hoping Exercise
- Core Stability Exercises (Experimental)
  Interventions: Other: Core Stability Exercises

INTERVENTIONS:
Other: Hoping Exercise — Week 1 Hopping to the sides on two legs (hands-free) 3 × 10 repetitions Hopping to front and back on two legs (hands-free) 3 × 10 repetitions Hopping to the front on two legs (hands-free) 3 × 10 repetitions Week 2 Hopping to the sides on two legs (hands on the chest) 2 × 15 repetitions Hopping to front and back on two legs (hands-free) 2 × 10 repetitions Hopping to the sides on one leg (hands-free) 5 × 4 repetitions Week 3 Hopping to the sides on one leg (hands on the chest) 3 × 10 repetitions Hopping zig-zag on two legs (hands-free) 2 × 10 repetitions Week 4 Hopping zig-zag on one leg (hands-free) 2 × 10 repetitions Hopping through squares on two legs (hands-free) 2 × 10 repetitions Week 5 Hopping in 8-shape on two legs (hands-free) 2 × 10 repetitions Hopping through squares on one leg (hands-free) 2 × 10 repetitions Week 6 Hopping through squares on one leg (hands on the chest) 2 × 10 repetitions Hopping in 8-shape on one leg (hands-free) 2 × 10 repetitions
  Arms: Hoping Exercise
Other: Core Stability Exercises — Week 1 Bridging in face-down position 3 × 20 s Bridging in the supine position 3 × 20 s Side bridging (right and left) 3 × 20 s Week 2 Lifting the leg in supine position (knee bent) 3 × 20 repetitions Rising opposite hand and foot in quadriceps 3 × 20 repetitions Cross-crunch abdominal muscles 3 × 20 repetitions Week 3 Bridging on a physioball 3 × 20 repetitions Cobra exercise on a physioball 3 × 20 repetitions Superman exercise 3 × 20 repetitions Week 4 Sit-up on a physioball 3 × 20 repetitions Rotating the trunk in a sitting position using a physioball 3 × 20 repetitions Week 5 Lunge exercise with trunk rotation using a medicine ball 3 × 20 repetitions Bridging on a physioball (leg raising alternately) 3 × 10 repetitions on each leg Week 6 Lunge exercise (back leg on a physioball) 3 × 10 repetitions on each leg Superman exercise (alternately) 3 × 10 repetitions on each side
  Arms: Core Stability Exercises

SUMMARY:
comparative effects of core versus hoping exercises on trunk stability and balance among kabaddi athlets

DETAILED DESCRIPTION:
Comparative effects of core stability exercises versus hopping exercises on trunk stability and balance among kabaddi athletes

ELIGIBILITY:
Inclusion Criteria:

* Males
* Aged 18-35 years
* Active players training for at least from 6 weeks
* Normal BMI (18.5-24.9 kg/m2)

Exclusion Criteria:

* Any acute inflammatory conditions of the back, spinal fractures, and systemic conditions affecting muscle performance,
* Spinal instability or any musculoskeletal, cardiac issue
* Presence of neurological deficits: history of seizure, headache, spinal cord injury

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
⦁ Y balance test | 8 weeks
  The YBT for the UQ (UQYBT) is reliable for assessing unilateral UE function in a closed chain position. The UQYBT also has the patient reach three directions with one UE while in a push-up position. The LQYBT has the patient stand on one leg while reaching out in 3 different directions with the other lower extremity. They are anterior, posteromedial and posterolateral. When using the Y-Balance test kit, the 3 reaches yield a "composite reach distance" or composite score used to predict injury.(18)
⦁ Stork stands balance test to measure static and dynamic equilibrium | 8 wee
  The stork balance test requires the person to stand on one leg, up on the ball of the foot, for as long as possible. The total time in seconds is recorded. The score is the best of three attempts. The table lists general ratings for this test. The stork test determines athletes' strength, conditioning, and technique and is reliable as long as it is done consistently.(30)

CONTACTS AND LOCATIONS:
Overall Officials: Wajeeha Zia, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No